CLINICAL TRIAL: NCT03188237
Title: AfyaJamii (Parenting Well): Evaluating the Feasibility of a Group Antenatal and Well-child Care Model in Pregnancy in Kenya
Brief Title: AfyaJamii (Parenting Well): Evaluating the Feasibility of a Group Antenatal/Well-child Care Model in Pregnancy in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moi University (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Astrid Christoffersen-Deb, Visiting Lecturer, Moi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMoi2
Record Dates: First submitted 2017-05-31; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Pregnancy Related; Group, Peer

STUDY DESIGN:
Intervention Model Description: AfyaJamii is a group care model in pregnancy facilitated by Government of Kenya (GOK) Community Health Volunteers (CHVs) and Ministry of Health (MOH) nurses. Pregnant women are assigned to specific care groups according to their Expected Date of Delivery (EDD) and meet 3 times antenatally and 4 times postnatally. These groups are meant to provide women with antenatal and postnatal care, peer support, and knowledge to improve their health outcomes and the health outcomes of their infants. This model of group prenatal and postnatal care is being evaluated as an alternative to the existing policy of focused antenatal care that individualizes care to a single woman at a time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AfyaJamii facility (Experimental): Facilities using AfyaJamii
  Interventions: Behavioral: AfyaJamii
- Referent facility (No Intervention): Facilities using Focused Antenatal Care Individual Model

INTERVENTIONS:
Behavioral: AfyaJamii — AfyaJamii is a group antenatal and well-child care program developed in Kenya for use in Kenyan health centers
  Arms: AfyaJamii facility

SUMMARY:
This proposal is a program evaluation of a group care delivery model designed for pregnant women that was implemented as a pilot project in Teso District, Kenya in 2012.

DETAILED DESCRIPTION:
The investigators will carry out a pre/post evaluation of this program comparing maternal and child health indicators collected at the facility and at 10 comparison facilities in the year prior to implementation (2012) and throughout the duration of the program (2013-2014). They will also analyze program attendance records, anonymous exit surveys, and training records.

ELIGIBILITY:
Inclusion Criteria:

* All facilities that participated in AfyaJamii

Exclusion Criteria:

* Any facility that did not offer AfyaJamii and was not been selected as a comparison facility

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Facility 4 Antenatal Care (ANC) visits | 18 months
  Average monthly number 4 or more ANC facility visits

SECONDARY OUTCOMES:
Facility New Family Planning (FP) | 18 months
  Average monthly number new FP visits
Facility Total FP | 18 months
  Average monthly number total FP visits
Facility Delivery Rate | 18 months
  Average monthly number of Facility deliveries
Facility Oral Polio Vaccine 0 (OPV0) | 18 months
  Average monthly number of OPV0 Immunization

CONTACTS AND LOCATIONS:
Overall Officials: Julia Songok, MBChB, Principal Investigator — Moi University
Locations (1):
- Teso North Ministry of Health Centers, Kocholya, Kenya

IPD SHARING:
Plan to Share IPD: No